CLINICAL TRIAL: NCT06522321
Title: Radiographic Assessment of Bone Dimension Around Immediate Implants With FDBA and I-PRF vs FDBA Alone- A Randomized Clinical Controlled Trial
Brief Title: Radiographic Assessment of Bone Dimension Around Immediate Implants With FDBA and I-PRF vs FDBA Alone
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, HOD OF PERIODONTOLOGY, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_147480
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Bone Density Increased
Keywords: Injectable platelet rich fibrin; bone dimensions; freeze dried bone allograft
MeSH Terms: conditions — Osteosclerosis | interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Intervention Model Description: Purposive Sampling technique will be done. All the patients who meet the eligibility criteria will be screened and then 20 patients will be randomly allotted into either of the two groups. The treatment allocation to the test and control group will be assigned by means of a sealed envelope containing a code derived from a computer-generated randomized list to receive either -
  1. TEST GROUP (n =10)- FDBA and PRF(i-prf) with immediate implant placement.
  2. CONTROL GROUP (n = 10) - FDBA alone with immediate implant placement.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiographic Assessment of Bone Dimension Around Immediate with FDBA and i-PRF vs FDBA (Experimental): TEST GROUP: FDBA and I-PRF with immediate implant placement. Local anesthesia is given. Atraumatic extraction is done. I-PRF is prepared by centrifugation procedure. Osteotomy is done at the selected site after radiographic assessment. Immediate implant is placement along with I-PRF and FDBA. Suture is placed at the surgical site.
  Interventions: Biological: i-PRF and FDBA
- Radiographic Assessment of Bone Dimensions Around Immediate Implants With FDBA and I-PRF vs FDBA (Experimental): CONTROL GROUP: FDBA alone with immediate implant placement. Local anesthesia is given. Atraumatic extraction is done.Osteotomy is done at the selected site after radiographic assessment. Immediate implant is placement along with FDBA alone. Suture is placed at the surgical site.
  Interventions: Biological: i-PRF and FDBA

INTERVENTIONS:
Biological: i-PRF and FDBA — A mucoperiosteal flap will be raised and atraumatic extraction will be done. An immediate implant with FDBA and I-PRF (experimental group) will be placed according to the standard protocol.
  An immediate implant with FDBA( comparative group) will be placed according to the standard protocol .
  The surgical wound closure will be coapted with sutures
  Other Names: platelet rich fibrin and freeze dried bone

SUMMARY:
The present study is a human, prospective, parallel, randomised controlled clinical trial conducted for radiographic assessment of bone dimension around immediate implants with FDBA and I-PRF vs FDBA Alone The trial is in accordance with the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010.

DETAILED DESCRIPTION:
Twenty healthy individuals satisfying the inclusion and exclusion criteria were recruited for the study. A detailed, thorough medical and dental history was obtained and each patient was subjected to comprehensive clinical and radiological examination. All patients were informed about the nature of the study, the surgical procedure involved, potential benefits and risks associated with the surgical procedure and written informed consent were obtained from all patients. All the patients were treated with immediate implants in endodontically and periodontically compromised sites. FDBA graft along with I-PRF is combined to form a sticky bone, this stable element is placed around the implants where bone is compromised.

The clinical and radiographic parameters were recorded at baseline, three months and six months postoperatively

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18-55 years of age.
2. Presence of non-restorable single rooted teeth (maxillary or mandibular) due to trauma, caries, root resorption, root fracture, endodontic or periodontal failure.
3. Grade I or Grade II extraction socket according to El Chaar et al 2016.
4. Good oral hygiene.
5. Good patient compliance.

Exclusion Criteria:

1. Systemic complications (uncontrolled diabetes and severe cardiovascular or infectious diseases).
2. Intravenous and oral bisphosphonate therapy.
3. Patients who are psychologically unable to participate.
4. Pregnant patients, patients with bone diseases and patients on chemotherapy or radiotherapy, alcohol or drug abuse.
5. Patients with hemorrhagic disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-08-25 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
Bone fill | At baseline, 3 months and 6 months
  Standard digital radiographs were taken at baseline, 3 months and 6 months by paralleling/long-cone technique. Radiographic images at all the time intervals were taken by using a metallic counting grid (IOPA film grid® , BlueDent, Chennai, India). The bone-fill was measured in square millimeters by point-counting the number of squares over newly developing radiopacities at different follow up periods. Squares that were half filled or unclear were not counted.
Bone dimensions | At baseline, 3 months and 6 months
  The sites will be assessed vertically and horizontally by CBCT images taken at baseline and 6 months after the implant placement.
Bone density | At baseline, 3 months and 6 months
  Bone mineral density is obtained by the CBCT (GENORAY (PAPAYA 3D premium operation software)
Marginal bone level | At baseline, 3 months and 6 months
  distance between reference point(the implant shoulder) and the first marginal bone-to-implant contact level using standard digital radiographs
Early wound healing index | At baseline, 3 months and 6 months
  SCORE 1: COMPLETE FLAP CLOSURE NO FIBRIN LINE IN THE INTERPROXIMAL AREA SCORE 2: COMPLETE FLAP CLOSURE FINE FIBRIN LINE IN THEINTERPROXIMAL AREA SCORE 3: COMPLETE FLAP CLOSURE FIBRIN CLOT IN THE INTERPROXIMAL AREA SCORE 4:INCOMPLETE FLAP CLOSURE PARTIAL NECROSIS OF THE INTERPROXIMAL AREA SCORE 5: INCOMPLETE FLAP CLOSURE COMPLETE NECROSIS OF THE INTERPROXIMAL AREA. SCORE 1: COMPLETE FLAP CLOSURE NO FIBRIN LINE IN THE INTERPROXIMAL AREA SCORE 2: COMPLETE FLAP CLOSURE FINE FIBRIN LINE IN THEINTERPROXIMAL AREA SCORE 3: COMPLETE FLAP CLOSURE FIBRIN CLOT IN THE INTERPROXIMAL AREA SCORE 4:INCOMPLETE FLAP CLOSURE PARTIAL NECROSIS OF THE INTERPROXIMAL AREA SCORE 5: INCOMPLETE FLAP CLOSURE COMPLETE NECROSIS OF THE INTERPROXIMAL AREA. Wachet et al wound healing index will be used for obtaining the healing index

SECONDARY OUTCOMES:
GINGIVAL INDEX | 3 months and 6 months
  The severity of gingivitis is scored on the mesiofacial and distofacial papillae, facial and lingual margin of selected teeth.
  A blunt instrument is used to assess the bleeding potential of tissues
  The index relies entirely on visual criteria of gingivitis and eliminates the use of probing or pressure to establish the presence or absence of bleeding.
GINIVAL BLEEDING INDEX | 3 months and 6 months
  The gingival bleeding index of Ainamo J and Bay I was developed as an easy and suitable way for assessing a patient's progress in Plaque control. The presence or absence of gingival bleeding is determined by gentle probing of the gingival crevice with a periodontal probe. The appearance of bleeding within 10 seconds indicates a positive score, which is expressed as percentage of the total number of gingival margin examined.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Prabhuji MLV, MDS, Study Chair — PROFESSOR AND HOD
Locations (1):
- Dr. Prabhuji MLV, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: No